CLINICAL TRIAL: NCT02986607
Title: Corticosteroid Rhythms in Hypoparathyroid Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Astor, MD, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/871
Record Dates: First submitted 2016-12-05; First posted 2016-12-08 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hypoparathyroidism; Hyperparathyroidism
MeSH Terms: conditions — Hypoparathyroidism; Hyperparathyroidism | interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypoparathyroidism (Experimental): Subcutaneous 24h microdialysis before PTH treatment and during continous subcutaneous PTH treatment. PTH, Natpara (parathyroid hormone 1-84) 50 µg doses with a concentration of 800 µg/ml, will be delivered by an insulin-pump (OmniPod) which delivers the infusion gear continous subcutaneously based on units (U) of insulin. 1 µg Natpara equals 0.125 U of infusion. The starting dose for pump treatment will be 0.50 µg per kilo per day and adjusted according to Calcium levels.
  Controls: patients With hyperparathyroidism and healthy volunteers will perform 24h microdialysis.
  Interventions: Drug: parathyroid hormon 1-84

INTERVENTIONS:
Drug: parathyroid hormon 1-84 — Hypoparathyroidism patients will receive Natpara in continous subcutaneous infusion delivered by a pump for 4-7 days.
  Other Names: Natpara

SUMMARY:
The investigators hypothesise that parathyroid hormon (PTH) depletion interferes with normal activity of the hypothalamus-pituitary-adrenal (HPA)-axis and the renin-angiotensin-aldosterone-system (RAAS), which in turn may impact morbidity and quality of life. The main objective of the current study is to test if PTH deficiency influences the secretion of corticosteroids and whether any abnormalities in the HPA-axis and the RAAS-system can be reversed by PTH infusion.

DETAILED DESCRIPTION:
Visit 1: Optimizing conventional treatment regarding s-magnesium, s-calcium, s-phosphorous and 25-hydroxyvitamin D (25(OH)D)-levels.

Visit 2 (In-hospital 4-7 days): Day one: 24h microdialysis sampling, venous blood sampling and 24h urine will be collected. Day 2: Start of PTH pump-treatment. Day 3-x: dose adjustment of PTH pump therapy according to Calcium Levels, the first two days after started PTH six daily venous blood-samplings will be performed. Day x: 24h microdialysis sampling and 24h urine-sampling and a venous blood sampling. Restart of conventional treatment.

The Control patients (healthy volunteers and patients with hyperparathyroidism) will perform 24h microdialysis-sampling only.

ELIGIBILITY:
Inclusion Criteria:

* Postsurgical hypoparathyroidism of at least one year duration. Undetectable PTH values (< 0.3 pmol/l) or less than 1.3 pmol/l despite hypocalcaemia (Reference range PTH: 1.3-6.8 pmol/L) must be documented before inclusion. 25-hydroxyvitamin D (25(OH)D) should be > 50 nmol/l prior to baseline.
* Healthy male and female volunteers, aged 18-60 years
* Patients with primary hyperparathyroidism, defined as simultaneous increased PTH and serum calcium levels, normal or increased urine calcium to exclude hypocalciuric hypercalcemia, normal kidney function (estimated glomerular filtration rate (eGFR) above 60), aged 18-60 years

Exclusion Criteria:

* Patients with diabetes mellitus, Addison's disease and patients on steroid medication will not be included in this study.
* Other exclusion criteria are unstable cardiovascular disease, active malignant disease, epilepsy, pregnancy or lactation, significant hepatic or kidney disease (alanine aminotransferase (ALAT) and or aspartate aminotransferase (ASAT) > 2 times upper limit of normal, eGFR < 30 ml/min), pharmacological treatment with PTH the last 3 months, treatment with other drugs that could interfere with interpretation of the results. Allergy to metacresol, lidocaine or multiple allergies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Corticosteroid secretion in hypoparathyroid patients | One week
  Evaluating of 24h corticosteroid secretion with PTH versus without PTH in hypoparathyroid patients with undetectable PTH-values

CONTACTS AND LOCATIONS:
Overall Officials: Eystein Husebye, Professor, Study Chair — UiB
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Astor MC, Lovas K, Methlie P, Simunkova K, Assmus J, Husebye ES. Corticosteroid rhythms in hypoparathyroid patients. Eur J Endocrinol. 2024 Aug 30;191(3):271-278. doi: 10.1093/ejendo/lvae102. PMID 39167533